CLINICAL TRIAL: NCT05528822
Title: Comparative Prospective Randomized Study of Modified Fascia Iliaca Compartment Block Versus Pericapsular Nerve Group Block in Elderly Patients' Total Hip Arthroplasty on the Post-operative Quality of Recovery
Brief Title: Study of H-FICB ＆ PENG Block in Elderly Patients' THA on the Post-operative Quality of Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-K090
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2022-09

CONDITIONS: Nerve Block; Quality of Recovery
Keywords: modified fascia iliaca compartment block; pericapsular nerve group block; the post-operative quality of recovery; HHS score; VAS score
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group F: H-FICB under ultrasound guidance before general anesthesia (Experimental): Group F was subjected to a high fascia iliaca compartment block under ultrasound guidance before general anesthesia.
  Interventions: Procedure: ultrasound-guided high fascia iliaca compartment block
- Group P: PENG block under ultrasound guidance before general anesthesia (Experimental): Group P was subjected to a pericapsular nerve group (PENG) Block under ultrasound guidance before general anesthesia.
  Interventions: Procedure: ultrasound-guided pericapsular nerve group (PENG) block

INTERVENTIONS:
Procedure: ultrasound-guided high fascia iliaca compartment block — H-FICB was guided by ultrasound before general anesthesia. The patient was supine. First, the probe is placed transversely above the groin. Then slide the probe up and down to reveal a clear image of the internal oblique and sartorius muscles. There is a bowtie-like iliac fascia space at the junction of these two muscles. After the scanning, the needle was inserted behind the probe with the tip pointed to the ventral side under the guidance of real-time ultrasound; the tip passed through the skin into the iliac fascia space and advanced to the inguinal ligament. After no blood was extracted, 1 ~ 2 ml of normal saline was firstly injected to determine whether the tip position was correct. If the needle tip was correctly positioned, 0.375% ropivacaine 30 mL of local anesthetic was injected. The H-FICB was performed under ultrasound guidance by the same anesthesiologist.
  Arms: Group F: H-FICB under ultrasound guidance before general anesthesia
Procedure: ultrasound-guided pericapsular nerve group (PENG) block — A low-frequency curvilinear transducer was placed in the transverse plane over the anterior inferior iliac spine (AIIS) and moved over inferiorly to visualize the pubic ramus. The femoral artery and ilio pubic eminence (IPE) were then visualized (Figure 1). Using in-plane technique 10 cm echogenic 21 gauge needle was advanced from lateral to medial direction, and 20 ml of local anesthetic 0.5% ropivacaine was deposited between the psoas tendon anteriorly and pubic ramus posteriorly.
  Arms: Group P: PENG block under ultrasound guidance before general anesthesia

SUMMARY:
Total joint replacement is projected to become the most common elective surgical procedure in the coming decade; the prevalence of total hip arthroplasty (THA) was estimated as more than 2.5 million individuals in the entire United States population. Orthopedic procedures involving the hip have remained challenging for regional anesthesia given the complex innervation, painful nature contributing to difficulty positioning, and a desire to maintain mobility to hasten postoperative recovery.

DETAILED DESCRIPTION:
By comparing the intraoperative and postoperative rehabilitation indexes of high fascia iliac nerve block and hip pericapsular nerve block, we can choose a more suitable analgesic method for this operation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 to 80 years male and female
* Scheduled for elective single-incision laparoscopic cholecystectomy
* The patients volunteered to participate in the study and signed the informed consent

Exclusion Criteria:

* Preexisting neuropathy
* Coagulopathy
* Local skin infection
* Hepatic, renal or cardiorespiratory failure
* Local anesthetic allergy
* Pregnancy
* Complications of gallstone with gallbladder perforation
* Diffuse peritonitis
* Acute pyogenic cholangitis

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline visual analogue scale | one day before the operation.
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0 to 100. A higher score indicates greater pain intensity. Based on the distribution of pain Visual Analogue Scale scores in post-surgical patients (knee replacement, hysterectomy, or laparoscopic myomectomy) who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain Visual Analogue Scale have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Harris Hip Score | At one week, one month, and three months post-operatively.
  The HHS is divided into three sections. The first section are questions about pain and its impact which are answered by the patient or client. The second and third sections require the physiotherapist to assess the patient or client's hip joint and function.The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. Results can be recorded and calculated online. The maximum score possible is 100. Results can be interpreted with the following[1]: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.

SECONDARY OUTCOMES:
The mini-mental State Examination | one day before the operation.
  The mini-mental State Examination is effective as a screening tool for cognitive impairment in older, community-dwelling, hospitalized, and institutionalized adults. Assessment of an older adult's cognitive function is best achieved when it is done routinely, systematically, and thoroughly. The Mini-Mental State Examination (MMSE) or Folstein test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. Any score of 24 or more (out of 30) indicates normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points), or mild (19-23 points) cognitive impairment. The raw score may also need to be corrected for educational attainment and age.

CONTACTS AND LOCATIONS:
Overall Officials: Xingguo Xu, Principal Investigator — Chair
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No